CLINICAL TRIAL: NCT02107625
Title: A Multi-centre, Randomized, Single-blind, Comparative Trial: Traditional Dietary Advice Versus a Low FODMAP Diet Intake in IBS Patients
Brief Title: Traditional Dietary Advice Versus a Low FODMAP Diet Intake in IBS Patients
Acronym: KRIBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Karolinska Institutet (Other); Aleris Specialistvård Sabbatsberg (Unknown)
Responsible Party: Principal Investigator, Hans Törnblom, MD, PhD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KRIBS1
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Irritable Bowel Syndrome
Keywords: Defecation; Abdominal pain
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet A i.e. Low FODMAP diet (Experimental): The patients are thoroughly informed verbally and in writing how to eat according to the low FODMAP diet. The diet imply restrictions in carbohydrate intake and the patients need to follow a list with yes/no-foods for 4 weeks.
  Interventions: Behavioral: Diet A i.e. Low FODMAP diet
- Diet B, i.e. Traditional IBS diet (Experimental): The patients are thoroughly informed verbally and in writing how to eat according to traditional IBS dietary advices. The diet imply adapting to regular dietary habit with meals 6 times a day, no to big meals, to chew food thoroughly, to peel fruits and vegetables, no carbonated beverages, no chewing gum, no soft drinks, no sugar-free candies, or cookies. Reduce spicy foods, coffee, alcohol, onion, pulses, and fatty foods. Keep strictly to the dietary advice for 4 weeks.
  Interventions: Behavioral: Diet B, i.e. Traditional IBS diet

INTERVENTIONS:
Behavioral: Diet A i.e. Low FODMAP diet
  Arms: Diet A i.e. Low FODMAP diet
Behavioral: Diet B, i.e. Traditional IBS diet
  Arms: Diet B, i.e. Traditional IBS diet

SUMMARY:
The purpose of this study is to to assess if the new diet with a low-FODMAP(Fermented Oligo-, Di-, Monosaccharides And Polyols) -content yields a milder symptom picture in IBS patients compared to traditionally dietary advice in IBS. The study also aim to investigate patients compliance to either dietary advices. Further, the investigators aim to find out if IBS patients with different symptoms are alleviated in different ways, to be able to individualize the dietary advices to result in a more optimal symptom relief in each patient in the future.

ELIGIBILITY:
Inclusion Criteria:

* IBS diagnosis
* Adult (over 18 years)
* Be able to read/understand/write swedish

Exclusion Criteria:

* Severe heart failure
* Severe liver disease
* Severe neurologic disease
* Severe psychological disease
* Severe gastrointestinal disease (i.e. celiac disease, IBD (inflammatory bowel disease) e.g.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Symptom alleviation through the questionnaire IBS-SSS | 4 weeks
  IBS-SSS i.e. the IBS Severity Scoring System. To assess the possible change of severity of IBS symptoms. The overall IBS score is calculated ranging from 0 to 500. A higher score implicates more severe symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Törnblom, MD, PhD, Principal Investigator — Sahlgrenska University Hospital

REFERENCES:
- [Derived] Nybacka S, Colomier E, Pall Hreinsson J, Storsrud S, Tack J, Tornblom H, Simren M. Dietary Intake and Quality in Irritable Bowel Syndrome: A Comparative Study With Controls and the Association With Symptom Severity. Am J Gastroenterol. 2024 Nov 27;120(9):2154-2164. doi: 10.14309/ajg.0000000000003249. PMID 39601420
- [Derived] Nybacka S, Simren M, Storsrud S, Tornblom H, Winkvist A, Lindqvist HM. Changes in serum and urinary metabolomic profile after a dietary intervention in patients with irritable bowel syndrome. PLoS One. 2021 Oct 11;16(10):e0257331. doi: 10.1371/journal.pone.0257331. eCollection 2021. PMID 34634050
- [Derived] Nybacka S, Storsrud S, Liljebo T, Le Neve B, Tornblom H, Simren M, Winkvist A. Within- and Between-Subject Variation in Dietary Intake of Fermentable Oligo-, Di-, Monosaccharides, and Polyols Among Patients with Irritable Bowel Syndrome. Curr Dev Nutr. 2018 Dec 24;3(2):nzy101. doi: 10.1093/cdn/nzy101. eCollection 2019 Feb. PMID 30838348
- [Derived] Bennet SMP, Bohn L, Storsrud S, Liljebo T, Collin L, Lindfors P, Tornblom H, Ohman L, Simren M. Multivariate modelling of faecal bacterial profiles of patients with IBS predicts responsiveness to a diet low in FODMAPs. Gut. 2018 May;67(5):872-881. doi: 10.1136/gutjnl-2016-313128. Epub 2017 Apr 17. PMID 28416515
- [Derived] Bohn L, Storsrud S, Liljebo T, Collin L, Lindfors P, Tornblom H, Simren M. Diet low in FODMAPs reduces symptoms of irritable bowel syndrome as well as traditional dietary advice: a randomized controlled trial. Gastroenterology. 2015 Nov;149(6):1399-1407.e2. doi: 10.1053/j.gastro.2015.07.054. Epub 2015 Aug 5. PMID 26255043